CLINICAL TRIAL: NCT06138678
Title: Vastra Gotaland Region Accelerated Transcranial Magnetic Stimulation Treatment for Depression
Brief Title: VGR Accelerated TMS Treatment for Depression
Acronym: VAiT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other); Uppsala University (Other); The Swedish Society of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAiT
Record Dates: First submitted 2023-10-27; First posted 2023-11-18 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Depression
Keywords: iTBS; rTMS; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Accelerated iTBS protocol (Experimental): Magnetic pulses of 120% of visual motor threshold applied in triplets of 50 Hz bursts, repeated at 5 Hz; 2 seconds on and 8 seconds off; 1200 pulses per session; total duration of 6 min 40 s over the left DLPFC (F3), given in 2 sessions per day (50 min interval) on 15 week days.
  Interventions: Device: iTBS (intermittent theta-burst stimulation)
- Routine iTBS protocol (Active Comparator): Magnetic pulses of 120% of visual motor threshold applied in triplets of 50 Hz bursts, repeated at 5 Hz; 2 seconds on and 8 seconds off; 600 pulses per session; total duration of 3 min 20 s over the left DLPFC (F3), given in 1 session per day on 30 week days.
  Interventions: Device: iTBS (intermittent theta-burst stimulation)

INTERVENTIONS:
Device: iTBS (intermittent theta-burst stimulation) — The iTBS treatment is a type of rTMS (repetitive transcranial magnetic stimulation), delivered with MagPro R30 stimulator and a conventional cool-B65 coil.
  The iTBS treatment is applied to over the dorsolateral prefrontal cortex using a standardized measuring of the anatomical landmark F3 from the 10-20 positioning system. The coil is positioned with the handle at in a 45 degree angle from the midline. The centre of the butterfly is placed towards the patient head.

SUMMARY:
Intermittent theta burst stimulation (iTBS), a variant of repetitive transcranial magnetic stimulation (rTMS), is a well documented method for treatment of depression.

The aim of the study is to assess the effect of an accelerated iTBS protocol compared to a routine iTBS protocol. In the accelerated protocol patients will receive 1200 pulses per session (2 sessions per day, 15 treatment days) and in the routine protocol patients will receive 600 pulses per session (1 session per day, 30 treatment days).

Participants (n = 146) will be recruited among patients referred to iTBS and randomized to treatment. Participants will be assessed by a psychiatrist, or a resident psychiatrist, prior to treatment to assure that they fulfill all inclusion criteria and non of the exclusion criteria. A psychiatrist, or a resident psychiatrist, will assess depressive symptoms 3 and 6 weeks after first day of treatment. Patients will complete self-rating questionnaires during screening, weekly for 6 weeks starting from the first day of treatment, and 6 months after end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of depression verified through a Mini International Neuropsychiatric Interview (M.I.N.I.)
* MADRS-S >= 20
* unchanged medication last month
* unchanged psychological treatment last month
* admitted to psychiatric ward last month
* no ECT or TMS last six months
* provision of signed informed consent form
* indication for TMS is depression

Exclusion Criteria:

* addiction (illicit drugs or alcohol)
* pregnancy
* epilepsy
* conductive ferromagnetic or other metals implanted in the head or within 30 cm of the treatment coil
* implanted device that is activated or controlled in any way by physiological signals
* implanted mediation pumps
* intracardiac lines, even when removed
* regular use of benzodiazepines
* any condition that seriously increases the risk of non-compliance or loss of follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Difference in MADRS-S from baseline to three weeks after first iTBS treatment | 3 weeks
  The self-rating version of the Montgomery-Asberg Depression Rating Scale (MADRS-S) is a rating scale (0-54 points), where a higher score indicates worse depressive symptoms

SECONDARY OUTCOMES:
Difference in MADRS-S from baseline to one week after first iTBS treatment | 1 week
  The self-rating version of the Montgomery-Asberg Depression Rating Scale (MADRS-S) is a rating scale (0-54 points), where a higher score indicates worse depressive symptoms
Difference in MADRS-S from baseline to two weeks after first iTBS treatment | 2 weeks
  The self-rating version of the Montgomery-Asberg Depression Rating Scale (MADRS-S) is a rating scale (0-54 points), where a higher score indicates worse depressive symptoms
Difference in MADRS-S from baseline to four weeks after first iTBS treatment | 4 weeks
  The self-rating version of the Montgomery-Asberg Depression Rating Scale (MADRS-S) is a rating scale (0-54 points), where a higher score indicates worse depressive symptoms
Difference in MADRS-S from baseline to five weeks after first iTBS treatment | 5 weeks
  The self-rating version of the Montgomery-Asberg Depression Rating Scale (MADRS-S) is a rating scale (0-54 points), where a higher score indicates worse depressive symptoms
Difference in MADRS-S from baseline to six weeks after first iTBS treatment | 6 weeks
  The self-rating version of the Montgomery-Asberg Depression Rating Scale (MADRS-S) is a rating scale (0-54 points), where a higher score indicates worse depressive symptoms
Difference in MADRS-S from baseline to six months after last iTBS treatment | 6 months
  The self-rating version of the Montgomery-Asberg Depression Rating Scale (MADRS-S) is a rating scale (0-54 points), where a higher score indicates worse depressive symptoms
Difference in QIDS-SR from baseline to one week after first iTBS treatment | 1 week
  The self-rating Quick Inventory of Depressive Symptomatology (QIDS-SR) is a rating scale (0-27 points), where a higher score indicates worse depressive symptoms
Difference in QIDS-SR from baseline to two weeks after first iTBS treatment | 2 weeks
  The self-rating Quick Inventory of Depressive Symptomatology (QIDS-SR) is a rating scale (0-27 points), where a higher score indicates worse depressive symptoms
Difference in QIDS-SR from baseline to three weeks after first iTBS treatment | 3 weeks
  The self-rating Quick Inventory of Depressive Symptomatology (QIDS-SR) is a rating scale (0-27 points), where a higher score indicates worse depressive symptoms
Difference in QIDS-SR from baseline to four weeks after first iTBS treatment | 4 weeks
  The self-rating Quick Inventory of Depressive Symptomatology (QIDS-SR) is a rating scale (0-27 points), where a higher score indicates worse depressive symptoms
Difference in QIDS-SR from baseline to five weeks after first iTBS treatment | 5 weeks
  The self-rating Quick Inventory of Depressive Symptomatology (QIDS-SR) is a rating scale (0-27 points), where a higher score indicates worse depressive symptoms
Difference in QIDS-SR from baseline to six weeks after first iTBS treatment | 6 weeks
  The self-rating Quick Inventory of Depressive Symptomatology (QIDS-SR) is a rating scale (0-27 points), where a higher score indicates worse depressive symptoms
Difference in QIDS-SR from baseline to six months after first iTBS treatment | 6 months
  The self-rating Quick Inventory of Depressive Symptomatology (QIDS-SR) is a rating scale (0-27 points), where a higher score indicates worse depressive symptoms
Difference in SDS from baseline to six weeks after first iTBS treatment | 6 weeks
  The Sheehan Disability Scale (SDS) is a self-rating assessment (0-30 points), where a higher score indicates more pronounced functional impairment
Difference in SDS from baseline to six months after first iTBS treatment | 6 months
  The Sheehan Disability Scale (SDS) is a self-rating assessment (0-30 points), where a higher score indicates more pronounced functional impairment
Difference in EQ-VAS from baseline to three weeks after first iTBS treatment | 3 weeks
  The EQ-5D visual analogue scale (EQ-VAS) is a self-rating assessment (VAS 0-100 points), where a higher (VAS) score indicates a higher health-related quality of life
Difference in EQ-VAS from baseline to six weeks after first iTBS treatment | 6 weeks
  The EQ-5D visual analogue scale (EQ-VAS) is a self-rating assessment (VAS 0-100 points), where a higher (VAS) score indicates a higher health-related quality of life
Difference in EQ-VAS from baseline to six months after first iTBS treatment | 6 months
  The EQ-5D visual analogue scale (EQ-VAS) is a self-rating assessment (VAS 0-100 points), where a higher (VAS) score indicates a higher health-related quality of life
Difference in CGI-S from baseline to three weeks after first iTBS treatment | 3 weeks
  The Clinical Global Impression - Severity scale (CGI-S) is a clinical rating scale (0-7 points), where a higher score indicates more severe symptoms
Difference in CGI-S from baseline to six weeks after first iTBS treatment | 6 weeks
  The Clinical Global Impression - Severity scale (CGI-S) is a clinical rating scale (0-7 points), where a higher score indicates more severe symptoms
Difference in CGI-I from baseline to three weeks after first iTBS treatment | 3 weeks
  The Clinical Global Impression - Improvement scale (CGI-I) is a clinical rating scale (0-7 points) of symptom improvement (lower score)/worsening (higher score) compared to baseline
Difference in CGI-I from baseline to six weeks after first iTBS treatment | 6 weeks
  The Clinical Global Impression - Improvement scale (CGI-I) is a clinical rating scale (0-7 points) of symptom improvement (lower score)/worsening (higher score) compared to baseline
Number of patients in remission three weeks after first iTBS treatment | 3 weeks
  A patient with a MADRS-S score of < 10 is considered to be in remission
Number of patients in remission six weeks after first iTBS treatment | 6 weeks
  A patient with a MADRS-S score of < 10 is considered to be in remission

CONTACTS AND LOCATIONS:
Overall Officials: Melker Hagsäter, MD, MSc, PhD, Principal Investigator — Västra Götaland Regional Council
Locations (2):
- Sweden (2):
  - Kungälv Hospital, Kungälv
  - Hospital of Skövde, Skövde

IPD SHARING:
Plan to Share IPD: No